CLINICAL TRIAL: NCT03760692
Title: Comparison of I-gel and Ambu AuraGain Without Neuromuscular Blocker in Laparoscopic Gynecological Surgery
Brief Title: I-gel vs Ambu AuraGain in Laparoscopic Gynecological Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Sule Ozbilgin, Director, Dokuz Eylul University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 351-SBKAEK; HUSE 012-ANR-2017 (Other: Hospital Universitario del Sureste)
Record Dates: First submitted 2018-11-27; First posted 2018-11-30 (Actual); Last update posted 2022-03-28 (Actual); Status verified 2022-03

CONDITIONS: Airway Morbidity; Anesthesia
Keywords: supraglottic airway device; laparoscopic gynecological surgery

STUDY DESIGN:
Intervention Model Description: Prospective, multicenter, randomized
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group i-gel (Active Comparator): Insertion of the airway device. The size of the airway device used is based on the manufacturers' recommendations and evaluation of its clinical performance
  Interventions: Device: i-gel
- Group Ambu Auragain (Experimental): Insertion of the airway device. The size of the airway device used is based on the manufacturers' recommendations and evaluation of its clinical performance
  Interventions: Device: Ambu AuroGain

INTERVENTIONS:
Device: i-gel — Evaluation of clinical performance in terms of insertion, ventilation and complications
  Other Names: Group i-gel
  Arms: Group i-gel
Device: Ambu AuroGain — Evaluation of clinical performance in terms of insertion, ventilation and complications
  Other Names: Group Ambu AuroGain
  Arms: Group Ambu Auragain

SUMMARY:
To compare the effects of i-gel and Ambu AuraGain on ventilation parameters and surgical view during Trendelenburg position laparoscopic gynecological surgery in cases administered positive pressure ventilation without the use of neuromuscular agents.

DETAILED DESCRIPTION:
Prospective, multicenter, randomized and double-blind study, aged from 18 to 65 years undergoing elective laparoscopic gynecological surgery.

The patients are randomly assigned to 2 groups:

Group i-gel Group Ambu AuraGain

Procedure:

The investigation protocol contains the following sections:

1. Induction of anaesthesia. For preoperative sedation 0.02 mg/kg midazolam IV will be administered. 2 minutes of 0.2 µ/kg/min remifentanil and 6 mg kg st-1 propofol infusion, IV 1-2 mg kg-1 propofol . No muscle relaxant will be used for insertion of the airway device.
2. Bispectral index values will be held between 40-60.Bispectral index values will be within this interval by increasing or decreasing propofol infusion by 1 mg/kg after additional bolus dose of propofol (1 mg/kg).
3. Insertion of the airway device. The size of the airway device used is based on the manufacturers' recommendations.
4. Anesthesia maintenance will be ensured by 50% O2/air with 0.1-0.4 µ kg/min-1 remifentanil and 4-10 mg/kg/hr propofol IV infusion
5. Functionality of the gastric drainage channel of the airway device
6. Measurement of airway seal pressure (oropharyngeal leak pressure (OLP): at baseline, and at 2 minutes after airway device insertion (T1), 10 minutes after insufflation (T2), before desufflation (T3), before removal of airway device (T4). The maximum pressure allowed is 40 cm H2O.
7. Ventilatory mechanics and parameters and hemodynamic parameters are measured at baseline, and at T1, T2, T3 and T4.
8. Perioperative complications: Cough, vomiting, laryngeal spasm, laryngeal Stridor, airway intervention requirements, hypoxia (SpO2 < 92%)
9. Removal of the airway device: Presence of blood - 3 level grading (1:no blood; 2: trace amounts of blood; 3: clear amounts of blood). Complications: sore throat ( VAS:10-point scale), dysphonia (yes/no), dysphagia (yes/no).

ELIGIBILITY:
Inclusion Criteria:

* ASA classification I-II
* Between 18-65 years
* Undergoing elective laparoscopic gynecological surgery

Exclusion Criteria:

1. Those with any neck or upper respiratory tract pathology
2. Those at risk of gastric content regurgitation/aspiration (previous upper GIS surgery, known hiatus hernia, gastroesophageal reflux, history of peptic ulcers, full stomach, pregnancy)
3. Those with low pulmonary compliance or high airway resistance (chronic pulmonary diseases)
4. Obese patients (BMI >35)
5. Those with throat pain, dysphagia and dysphonia
6. Those with possible or previous difficult airway
7. Those with operations planned for longer than 4 hours
8. Conversion to laparotomy
9. Neuromuscular blocking agent used

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2018-11-01 (Actual); Primary Completion 2024-11-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Insertion time | intraoperative
  The time taken to successfully place the device in seconds
Change in airway seal pressure | intraoperative
  The maximum oropharyngeal leak pressure attained for each device.

SECONDARY OUTCOMES:
Number of attempts at insertion | intraoperative
  The number of repeated attempts required for successfully placing the device. Each device was given a chance of 3 attempts if still unsuccessful after 3 attempts another device was placed.

CONTACTS AND LOCATIONS:
Overall Officials: Sule Ozbilgin, MD, Study Director — Dokuz Eylul University, School of Medicine, Department of Anesthesiology and Intensive Care
Locations (2):
- Sureste University Hospital, Department of Anesthesiology and Critical Care, Madrid, Spain
- Dokuz Eylul University, School of Medicine, Department of Anesthesiology and Intensive Care, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided